CLINICAL TRIAL: NCT00210691
Title: Risperidone Depot (Microspheres) in the Treatment of Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of Long-acting Injectable Risperidone in the Treatment of Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004291
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; intramuscular injection; psychotropic agents; long-acting risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to document the long-term safety and tolerability of risperidone, formulated as a long-acting injectable, in the treatment of patients with schizophrenia or schizoaffective disorder; in addition, to evaluate the long-term effectiveness of long-acting risperidone and its effect on quality of life

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. This safety study is an extension of a randomized, double-blind, multicenter, parallel group study that investigates effectiveness and safety of risperidone injected intramuscularly in patients with schizophrenia or schizoaffective disorder. The present open-label study evaluates 3 different doses of a formulation of risperidone injected into the muscle at 2 week intervals for at least 1 year in patients with these conditions. Assessments of effectiveness include the Clinical Global Impression (CGI) overall severity of illness scale. Quality of life will be assessed by the SF-36 Health Survey. Safety evaluations include incidence of adverse events, physical examinations, and evaluations of the injection site, clinical laboratory tests, electrocardiograms (ECGs), and Extrapyramidal Symptom Rating Scale (ESRS), a scale assessing muscle tone, gain, and abnormal movements. Injections every 2 weeks for at least 1 year, beginning at 25milligrams[mg] and increasing to 50mg or 75mg (maximum dose). Dosages may be increased or decreased at investigator's discretion. During the first 3 weeks, risperidone tablets (2mg) once daily to supplement injectable risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the double-blind study (RIS-USA-121) or withdrawn from that study for safety reasons or due to worsening of condition as determined by results from the CGI
* diagnosis of schizophrenia or schizoaffective disorder according to criteria of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DMS IV)
* otherwise healthy on the basis of physical examination, medical history, electrocardiogram, blood biochemistry and hematology tests, and urinalysis.

Exclusion Criteria:

* Known intolerance, sensitivity, serious adverse events, or unresponsiveness to risperidone
* diagnosis of DMS IV Axis I condition other than schizophrenia or schizoaffective disorder
* diagnosis of substance abuse or dependence
* use of psychostimulants or an antipsychotic medication other than risperidone
* known disease of the central nervous system (stroke, Parkinson's Disease, Huntington's Disease, Alzheimer's Disease, cancer)
* pregnant or nursing females, or those lacking adequate contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 1999-12; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events; Injection site evaluation; Extrapyramidal Sympton Rating Scale (ESRS) results at each visit for at least 1 year; Clinical evaluations (physical exams, laboratory tests) will be conducted throughout trial

SECONDARY OUTCOMES:
Clinical Global Impression Severity of illness subscale (CGI-Severity) at each visit for at least 1 year. SF-36 assessed yearly.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.